CLINICAL TRIAL: NCT02902328
Title: Accuracy Evaluation for Software-based Visualization of Anatomical Brain Structures Using Surgical Information Sciences Inc. Algorithms
Brief Title: Accuracy Evaluation for SIS Software-based Visualization of Anatomical Brain Structures
Status: Completed | Type: Observational
Sponsor: Surgical Information Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SurgicalIS
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Software Evaluation for Visualizing Anatomical Structures That Are Not Typically Identified on Clinical MR Images

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI data collection: A group of 30 subjects will be scanned on a 3 Tesla (T) and on a 7T MRI scanners. The images will be compared.

SUMMARY:
SIS has developed a software technology, based on machine learning and image processing, designed to enhance standard clinical images for the visualization of anatomical structures.

DETAILED DESCRIPTION:
A cohort of 30 subjects will be scanned on a clinical MRI scanner as well as on a 7 Tesla (T) scanner. Images acquired on the 7T allow to visualize anatomical structures that are not easily identified on standard clinical images.

SIS software will be used to visualize selected anatomical features on the clinical image and the results will be compared with the images of the same subject obtained from the 7T MRI.

ELIGIBILITY:
Inclusion Criteria:

* all subject that are willing to be scanned on a 3T and 7T MRI scanners and are not excluded by the exclusion criteria below.

Exclusion Criteria:

1. MRI exclusion criteria for 7T scans: presence of any metallic clip(s) or implantable medical devices (e.g., heart valve, aneurysm clip, coils or surgery, renal or aortic clips, shunts, stents or stent grafts, metal mesh/coil implants, neurostimulator, insulin pump, IVC filter, artificial knee or hip, metal plates, pins, screws or wires anywhere in the body, any other metal implants, etc.).
2. Pregnant women.
3. Subject under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 30 adults who will be scanned on a 3T and 7T MRI to obtain anatomical images of their brain.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Validation of the accurate visualization of brain structures based on SIS algorithms | one year

IPD SHARING:
Plan to Share IPD: No